CLINICAL TRIAL: NCT05294679
Title: Clinical Use of Ciprofol in Painless Colonoscopy: a Large Sample, Multicenter, Randomized, Double-blind, Parallel-controlled Clinical Study
Brief Title: Explore the Clinical Application Value of Ciprofol in Painless Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Mengchang Yang, Director, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GYSDYRMYY
Record Dates: First submitted 2022-02-17; First posted 2022-03-24 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Induction of Anaesthesia
Keywords: Propofol; Ciprofol
MeSH Terms: interventions — Propofol; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned 1:1 to receive intravenous ciprofol or propofol 1 hour before the start of treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, evaluation researchers and drug administration researchers were set up. The whole process of the experiment was blind not only to the subjects, but also to the evaluation researchers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Placebo Comparator): The initial dose of propofol was 2mg/kg, and the intravenous infusion time was 30s. Within 1 minute (inclusive) of the end of the initial dose: if the subject has achieved sufficient sedation (MOAA/S score =0), the colonoscopy will commence. If subjects' MOAA/S score ≥ 1 point, additional administration of cyclopofol will be allowed 1 minute after the end of the initial dose. If the MOAA/S score was 0 after 3 consecutive times of addition, sedation failure was determined, and the study was recorded and quit. The drug was given according to clinical needs and the examination was completed. Maintenance of sedation after colonoscopy: In order to maintain a certain degree of sedation after colonoscopy (MOAA/S score ≤1 point), the evaluator decides when to administer additional drugs.
  Additional administration of propofol: The additional dose was 0.5mg/kg/ time, and intravenous bolus was administered.
  Interventions: Drug: Propofol
- Ciprofol ground (Experimental): The initial dose of ciprofol was 0.4mg/kg, and the intravenous infusion time was 30s. Within 1 minute (inclusive) of the end of the initial dose: if the subject has achieved sufficient sedation (MOAA/S score =0), the colonoscopy will begin; If subjects' MOAA/S score ≥ 1 point, additional administration of ciprofol will be allowed 1 minute after the end of the initial dose. If the MOAA/S score was 0 after 3 consecutive times of addition, sedation failure was determined, and the study was recorded and quit. The drug was given according to clinical needs and the examination was completed. Maintenance of sedation after colonoscopy: In order to maintain a certain degree of sedation after colonoscopy (MOAA/S score ≤1 point), the evaluator decides when to administer additional drugs.
  Ciprofol supplemental administration: the supplemental dose was 0.1mg/kg/ time, and intravenous bolus was administered.
  Interventions: Drug: Ciprofol

INTERVENTIONS:
Drug: Propofol — All patients completed pre-anaesthesia assessment, signed informed consent, and completed vital signs on the day before surgery, with values as baseline vital signs. On the day of surgery, after routine preparation before colonoscopy (fasting for at least 6h and water restriction for at least 2h before surgery), venous access was established in the left hand. 0.5μg/kg fentanyl was administered intravenously after oxygen inhalation through a nasal catheter (4-6 L/min). About 3 minutes after fentanyl administration, sedation induction was performed with ciprofol or propofol immediately.
  Arms: Propofol group
Drug: Ciprofol — Ciprofol
  Arms: Ciprofol ground

SUMMARY:
This study used propofol as a positive control, and adopted a large-sample, multi-center, randomized, double-blind, positive parallel controlled trial design to explore the clinical application value of ciprofol in painless colonoscopy.

DETAILED DESCRIPTION:
Subjects were randomly assigned 1:1 to receive intravenous ciprofol or propofol 1 hour prior to diagnosis and treatment. A centralized random grouping method was used in this study. After screening subjects, the researchers in each test center will log in to the random system after being confirmed by the researchers of the center, fill in the screening information, obtain the random number information, and issue the corresponding study drugs according to the random number. Random shelter number was generated by SAS software, and was used as the total blind base pair drug number and imported into the centralized random grouping system. In this study, evaluation researchers and drug administration researchers were set up. The whole process of the experiment was blind not only to the subjects, but also to the evaluation researchers. Evaluation investigators and administration investigators were set up in this study. The administration investigators were only involved in the process of random grouping, drug dispensing and administration, and the other processes including informed consent of subjects, screening, evaluation of efficacy indicators and safety, and planned visits were all completed by the evaluation investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing painless colonoscopy;
2. Patients aged from 18 to 80 years old, no gender limitation; 3, 18 < BMI < 30kg/m2 [BMI = weight (kg)/ height (m) squared]

4. American Society of Anesthesiologists (ASA) grades ⅰ ~ ⅲ

Exclusion Criteria:

1. Preoperative blood pressure >160/100 mmHG or < 80/50 mmHG.
2. Preoperative ecg suggested heart rate <50 times/min;
3. Acute respiratory tract infection with no cured history within 2 weeks;
4. People with serious metabolic diseases such as heart, brain, lung, liver, kidney and diabetes;
5. Predict people who may have or have had difficult airway;
6. Patients with obvious electrolyte disorders such as hyperkalemia;
7. Long-term use of immunosuppressants such as hormones or history of adrenocortical inhibition;
8. People who are known to be allergic to emulsions and opioids;
9. Preoperative combined use of other sedative and analgesic drugs
10. Suspected abuse of narcotic analgesics or sedatives; 11, there are neuromuscular system diseases, mental diseases and other people do not cooperate with the communication;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
the incidence of hypotension | Day 1
  Perioperative hypotension was defined as systolic blood pressure below 90mmHg, diastolic blood pressure below 50mmHg, or systolic blood pressure below baseline

SECONDARY OUTCOMES:
the successful sedation time | Day 1
  When the Patients'MOAA/S was 0 as the successful sedation time
Blood pressure | Day 1
  Record the blood pressure at entering the room (T0) , after anesthesia administration (T1),at time points 2min after anesthesia administration (T2), 4min after anesthesia administration (T3), at the end of surgery (T4), 5min after surgery (T5), 10min after surgery (T6), and before leaving the chamber (T7)
Heart rate | Day 1
  Record the heart rate at entering the room (T0) , after anesthesia administration (T1),at time points 2min after anesthesia administration (T2), 4min after anesthesia administration (T3), at the end of surgery (T4), 5min after surgery (T5), 10min after surgery (T6), and before leaving the chamber (T7)
Respiratory rate | Day 1
  Record the respiratory rate at entering the room (T0) , after anesthesia administration (T1),at time points 2min after anesthesia administration (T2), 4min after anesthesia administration (T3), at the end of surgery (T4), 5min after surgery (T5), 10min after surgery (T6), and before leaving the chamber (T7)
Oxygen saturation（SpO2 %） | Day 1
  Record the oxygen satuaition at entering the room (T0) , after anesthesia administration (T1),at time points 2min after anesthesia administration (T2), 4min after anesthesia administration (T3), at the end of surgery (T4), 5min after surgery (T5), 10min after surgery (T6), and before leaving the chamber (T7)
Steward wakefulness Score | Day 1
  Minimum value =0, maximum value =6, the higher the score, the higher the degree of wakefulness
Directional force score | Day 1
  Minimum value =0, maximum value =10, the higher the score, the higher the degree of directivity
Incidence of adverse events | Day 1
  including injection pain, intraoperative muscle fibrillation, hypoxemia, body movement, and postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Mengchang Yang, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No